CLINICAL TRIAL: NCT05261360
Title: A Phase II Trial to Investigate Clinical Efficacy of Autologous Synovial Fluid Mesenchymal Stem Cell-Derived Exosome Application in Patients With Degenerative Meniscal Injury
Brief Title: Clinical Efficacy of Exosome in Degenerative Meniscal Injury
Acronym: KNEEXO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ayla Eker Sariboyaci, Assoc. Prof. Dr., Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 56733164/203
Record Dates: First submitted 2021-11-01; First posted 2022-03-02 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Knee; Injury, Meniscus (Lateral) (Medial); Meniscus Tear; Meniscus Lesion; Meniscus; Degeneration; Meniscus; Laceration; Meniscus Injury, Tibial; Knee Injuries; Knee Pain Swelling; Arthralgia
Keywords: Meniscal injury; Exosome; Mesenchymal Stem Cell; Synovial Fluid; Regeneration
MeSH Terms: conditions — Wounds and Injuries; Lacerations; Tibial Meniscus Injuries; Knee Injuries; Arthralgia

STUDY DESIGN:
Intervention Model Description: The study was planned as three arms. One arm will be the control group, and the other two arms will be the experimental group. The control group defines the group that did not receive treatment. Those in the experimental group, who are the participants other than the control group, will occur in both experimental groups. SF-MSC (synovial fluid-derived mesenchymal stem cells) will be applied intraarticularly to the experimental group's right knee, and the experimental group's right knee will be included in the SF-MSC treatment group. SF-MSC-EX (synovial fluid-derived mesenchymal stem cells-derived exosomes) will be applied intraarticularly to the experimental group's left knee, and the experimental group's left knee will be included in the SF-MSC-EX treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SF-MSC-EX Treatment Group (Experimental group's left knees) (Experimental): The left knee will receive 1 million cells/kg SF-MSC-EX (Synovial fluid mesenchymal stem cell-derived exosome) by intra-articular injection method.
  Interventions: Drug: SF-MSC-EX
- SF-MSC Treatment Group (Experimental group's right knees) (Experimental): The right knee will receive 1 million cells/kg SF-MSC (Synovial fluid-derived mesenchymal stem cell) by intra-articular injection method.
  Interventions: Drug: SF-MSC
- Control Group (No Intervention): Participants who received no treatment were defined as the control group.

INTERVENTIONS:
Drug: SF-MSC-EX — Intra-articular administration of synovial fluid-derived mesenchymal stem cells-derived exosomes
  Other Names: Intraarticular Exosome Treatment
  Arms: SF-MSC-EX Treatment Group (Experimental group's left knees)
Drug: SF-MSC — Intra-articular administration of synovial fluid-derived mesenchymal stem cells
  Other Names: Intraarticular Stem Cell Treatment
  Arms: SF-MSC Treatment Group (Experimental group's right knees)

SUMMARY:
Comparison of intra-articular administration of synovial fluid-derived mesenchymal stem cells-derived exosomes with synovial fluid-derived mesenchymal stem cells on the same patient.

DETAILED DESCRIPTION:
Mesenchymal stem cell-derived exosomes will be developed and patented as an advanced technology platform as an autologous treatment protocol to repair damaged cartilage tissue. The fact that this treatment is obtained from an autologous source will significantly contribute to the literature in the field of personalized therapy (personalized medicine) and will pave the way for discoveries. Experiences from clinical trials may guide the use of MSC exosomes in other tissue and cell damaged pathologies and immune pathologies or chronic inflammatory diseases.

This study was supported by a grant (1004, 20AG031) from The Scientific and Technological Research Council of Turkey (TUBITAK).

ELIGIBILITY:
Inclusion Criteria:

* Accepting the Informed Consent Form
* Degenerative meniscus damage grade 1, 2 or 3 on MRI in both right and left knees, and also the patient does not want surgical treatment
* Patients with the same degenerative meniscus grade in both knees
* Patients with ongoing pain
* Patients without a history of malignancy
* Absence of signs of unstable meniscus tear such as snagging or locking
* Patients with stage 0, 1 or 2 gonarthrosis according to Kellgren-Lawrence gonarthrosis staging
* Patients without lower extremity malalignment

Exclusion Criteria:

* Patients whose treatment method was explained and who did not accept the method
* Patients outside the working-age range
* Congenital lesion
* Patients requiring surgical treatment (e.g. bucket handle tear and locked knee)
* Active inflammatory or connective tissue disease is thought to affect the patient's pain (eg lupus, rheumatoid arthritis, fibromyalgia)
* Local or systemic infection
* Pregnant or breastfeeding women
* Active endocrine disorder that may affect the assessment of patient's pain (eg, hypothyroidism, diabetes)
* Active neurological disorder that may affect the assessment of the patient's pain (eg, peripheral neuropathy, multiple sclerosis)
* Active heart disease
* Presence of a pacemaker
* Conditions where MR-I is contraindicated
* Patients with stage 3 or 4 gonarthrosis according to Kellgren-Lawrence gonarthrosis staging
* Patients with lower extremity malalignment
* Patients with signs of unstable meniscus tear such as snagging or locking

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Knee Functions | Up to 12th months
  The functional evaluation of the participants will be evaluated on the Tegner-Lysholm knee scoring scale. In Tegner-Lysholm knee scoring, examinations for the knee joint (Limp, support, pain, instability, locking, swelling, stair-climbing, and squatting) will be evaluated, and a maximum of 100 and a minimum of 0 points will be given. According to the evaluation, <65 points are interpreted as bad, 65-83 points as fair, 84-90 points as good, >90 points as excellent. Scores will be recorded by being examined before treatment and at the 6th, and 12th months after treatment. Knee functions of the control group will be evaluated simultaneously, and the effects of treatments on knee function will be determined.
Evaluation of Physical Activity | Up to 12th months
  The physical activity evaluation of the participants will be evaluated with the IPAQ (international physical activity questionnaire) short form. IPAQ short form will be evaluated and recorded before treatment and at the 6th, and 12th months after treatment. The control group's physical activity will be evaluated simultaneously, and the effects of treatments on physical activity will be determined.
Evaluation of Pain | Up to 12th months
  Pain assessment of the participants will be evaluated with VAS (Visual analog scale). The VAS will be evaluated and recorded before treatment and at the 6th, and 12th months after treatment. The physical activity of the control group will be evaluated simultaneously, and the effects of treatments on pain will be determined.
Evaluation of Radiological Images | Up to 12th months
  Participants will receive knee x-ray imaging and knee magnetic resonance imaging before treatment. The same radiological imaging will be performed at the 6th and 12th months after the treatment. At the same time, the same radiological imaging will be performed on the control group, and the effects of treatments on radiological imaging will be evaluated.
Evaluation of Cytokine Levels and Cytokine Genes Analyzes | Up to 12th months
  Before treatment and at the 6th and 12th months after treatment, cytokine levels (IL-10, IL-6, TNF-α, IL-8, IL-1β, IFN-ɣ, IL-2, IL-4, IL-13, MCP-1, VEGF) and gene analyzes (IL-10, IL-6, TNF-α, IL-8, IL-1β, IFN-ɣ, IL-2, IL-4, IL-13, MCP-1, IL-1ra, MIP-1b, CTGF, TGFβ3, BMP-2, BMP-4, IGF-1, IGF-2, PDGF, EGF, and VEGF genes) will be checked in the samples taken from the synovial fluid and blood. Samples will be taken from the control group along with the treatment group. In this way, the effects of treatments on cytokine levels will be evaluated.
Evaluation of Edema | Up to 12th months
  Edema in both knees will be measured using a tape measure by marking the midpoints of both patellae. Pre-treatment measurements will be recorded. Measurements of both knees will be recorded at 6 months and 12 months after treatment. The knees of the patients not receiving treatment will be measured simultaneously, and the changes will be compared.
Evaluation of Knee Joint Range of Motion | Up to 12th months
  The range of motion of both knees will be measured using the "Baseline Digital Absolute+Axis Goniometer." Knee extension measurements will be made with the patient in the supine position and flexion in the prone position. Pre-treatment measurements will be recorded. Post-treatment 6th and 12th-month measurements will also be recorded. Measurements of patients not receiving treatment will be recorded simultaneously, and changes will be compared.
Monitoring of treatment-related complications | Up to 12th months
  Adverse effects and complications will be observed in the treatment group, except for the expected local reactions (redness, swelling, bruising, etc.) after the application.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Eker Sarıboyacı, AssocProfDr., Study Chair — Cell Therapy and Stem Cell Production Application and Research Center (ESTEM); Onur Uysal, AssocProfDr., Study Director — Cell Therapy and Stem Cell Production Application and Research Center (ESTEM); Ulukan İnan, ProfDr., Principal Investigator — Eskisehir Osmangazi University Faculty of Medicine Department of Orthopedy and Traumatology
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Results will be reported after the completion of the study.

REFERENCES:
- [Background] Tegner Y, Lysholm J. Rating systems in the evaluation of knee ligament injuries. Clin Orthop Relat Res. 1985 Sep;(198):43-9. PMID 4028566
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Pan H, Zhang P, Zhang Z, Yang Q. Arthroscopic partial meniscectomy combined with medical exercise therapy versus isolated medical exercise therapy for degenerative meniscal tear: A meta-analysis of randomized controlled trials. Int J Surg. 2020 Jul;79:222-232. doi: 10.1016/j.ijsu.2020.05.035. Epub 2020 Jun 6. PMID 32522685